CLINICAL TRIAL: NCT01278914
Title: Phase I/II Trial of Vaccine Therapy With mRNA- Transfected Dendritic Cells in Patients With Androgen Resistant Metastatic Prostate Cancer
Brief Title: Trial of Vaccine Therapy With mRNA- Transfected Dendritic Cells in Patients With Androgen Resistant Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Svein Dueland, senior physician, Oslo University Hospital
Other Study IDs: DC Prostate
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Dendritic Cells (DC) prostate

SUMMARY:
PRIMARY OBJECTIVES:

Determination of safety and toxicity of vaccination with mRNA transfected DC (based on blood samples, and adverse events).

SECONDARY OBJECTIVES:

Determine immunological response to the vaccine (induction of specific T-cell response) and assessment of tumour response.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 45 years of age.
* Must have histologically confirmed adenocarcinoma of the prostate.
* Must have evidence of disease progression while on LHRH agonist, or orchiectomy, with or without an antiandrogen for advanced prostate cancer. All patients will be maintained on the hormone regimen throughout this protocol that they were receiving at the time of entry or recent progression. Increasing PSA in three subsequent analysis.
* Must be ambulatory with a ECOG performance score of <2
* Lab.values as following :ANC ( 1.5 x 109/L; platelets ( 100 x 109/L, Hb ( 9 g/dL (( 5.6 mmol/L). Creatinine ( 140 µmol/L (1.6 mg/dL); if borderline, the creatinine clearance ( 40 mL/min, Bilirubin < 20% above the upper limit of normal, ASAT and ALAT ( 2.5 the upper limit of normal. Albumin ( 2.5 g/L).
* Prior radiotherapy: a minimum of 4 weeks (8 weeks in case of extensive prior radiotherapy) must have elapsed between the end of the prior radiotherapy and entry into the protocol.
* Prior chemotherapy: a minimum of 4 weeks must have elapsed prior to entry in the study.
* If the patient has received strontium-89 and alpha-radin, at least three months must have elapsed prior to entry in the study.
* Informed consent and expected cooperation of the patients for the treatment and follow-up must be obtained and documented according to the ICH-GCP Guidelines.

Exclusion Criteria:

* History of prior malignancy other than prostate cancer, clinically evident within the 24 months preceding enrolment into the study, except curatively-treated basal cell or squamous cell carcinoma of the skin.
* Active infection requiring antibiotic therapy.
* Significant cardiac or other medical illness that would limit activity or survival, such as severe congestive heart failure, unstable angina, or serious cardiac arrhythmia.
* Autoimmune disease treated with steroid(s)
* History of asthma, anaphylaxis or other serious adverse reactions to vaccines.
* History of immunodeficiency or autoimmune disease such as rheumatoid arthritis, systemic lupus erythematosus, scleroderma, polymyositis/dermatomyositis, juvenile onset insulin dependent diabetes, or a vasculitic syndrome.
* Chemotherapy or other potentially immune-suppressive therapy that has been administered within 4 weeks prior to vaccination.
* Impending untreated spinal cord compression or urinary outlet obstruction.
* Any reason why, in the opinion of the investigator, the patient should not participate.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-02-01 (Actual); Primary Completion 2004-08-10 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo university Hospital, Oslo, Norway